CLINICAL TRIAL: NCT07141485
Title: Comparison of the PeDiAC Score and Intubation Difficulty Scale in Pediatric Patients Aged 0-5 Years Undergoing Tracheal Intubation With Videolaryngoscopy
Brief Title: Comparison of PeDiAC and the Intubation Difficulty Scale in Pediatric Patients Intubated With Videolaryngoscopy
Acronym: VIDEOPED
Status: Not yet recruiting | Type: Observational
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Sponsor
Other Study IDs: PEDIAC-VL-2025-GID
Record Dates: First submitted 2025-08-19; First posted 2025-08-26 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Videolaryngoscopy; Difficult Airway, Videolaryngoscopes; Airway Management Assessment; Pediatric Anesthesia
Keywords: Pediatric intubation; Difficult airway; PeDiAC; Intubation Difficulty Scale (IDS); Videolaryngoscopy; Modified Cormack-Lehane classification; Pediatric anesthesia; Tracheal intubation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pediatric Patients Undergoing Videolaryngoscopic Intubation: This group includes pediatric patients aged 0-5 years undergoing elective or emergency surgery under general anesthesia with videolaryngoscopic intubation. All patients will be evaluated for intubation difficulty using both the PeDiAC and the Intubation Difficulty Scale (IDS).

SUMMARY:
This prospective observational study aims to compare the effectiveness of the Paediatric Videolaryngoscopic Intubation and Difficult Airway Classification (PeDiAC) and the Intubation Difficulty Scale (IDS) in evaluating difficult tracheal intubation in pediatric patients aged 0 to 5 years. Patients undergoing general anesthesia with videolaryngoscopic intubation will be assessed using both scoring systems. The study seeks to determine which system more accurately reflects the difficulty of intubation and serves as a better guide for future anesthetic management, ultimately contributing to improved patient safety.

DETAILED DESCRIPTION:
This prospective observational study aims to compare the effectiveness of two scoring systems-Paediatric Videolaryngoscopic Intubation and Difficult Airway Classification (PeDiAC) and the Intubation Difficulty Scale (IDS)-in assessing the difficulty of tracheal intubation in pediatric patients aged 0 to 5 years. Pediatric patients undergoing elective or emergency surgery under general anesthesia will be included in the study. All intubations will be performed using a C-MAC videolaryngoscope.

Demographic data such as age, sex, weight, height, ASA physical status, and comorbidities will be recorded. Intraoperative monitoring parameters including peripheral oxygen saturation (SpO₂) and heart rate will also be documented. During intubation, the glottic view will be graded according to the Modified Cormack-Lehane classification.

Additional variables-including the time required to achieve optimal glottic visualization, total intubation time (from insertion of the device to cuff inflation), number of intubation attempts, and any complications (e.g., desaturation, mucosal bleeding)-will be noted.

Following intubation, both the intubating anesthesiologist and an independent observer will assign a subjective difficulty score using a visual analog scale ranging from 0 (extremely easy) to 10 (impossible). Subsequently, PeDiAC and IDS scores will be calculated for each case.

The primary objective is to determine which of the two scoring systems more accurately reflects the actual difficulty of tracheal intubation in this age group and to identify the one that may better guide future airway management strategies-ultimately aiming to improve safety and clinical outcomes in pediatric anesthesia.

ELIGIBILITY:
Eligible participants will be pediatric patients aged 0 to 5 years who are undergoing general anesthesia for any surgical procedure. All included patients must undergo tracheal intubation using a videolaryngoscope (C-MAC). Patients must have an ASA physical status classification of I to IV and written informed consent must be obtained from a parent or legal guardian prior to participation.

Inclusion Criteria:

* Pediatric patients between 0 and 5 years of age
* Undergoing general anesthesia for any type of surgical procedure
* ASA physical status classification I to IV
* Written informed consent obtained from parents or legal guardians

Exclusion Criteria:

* Patients undergoing awake fiberoptic intubation
* History of tracheal resection or reconstruction surgery
* Refusal to participate or absence of informed consent

Ages: 0 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: This study will enroll pediatric patients aged 0 to 5 years who are undergoing general anesthesia for elective and emergent surgical procedures requiring tracheal intubation. Patients will be intubated using a videolaryngoscope. Subjects with difficult airway history, emergency surgery, or airway pathology will be excluded. The study aims to compare two scoring systems evaluating intubation difficulty in this age group.
Sampling Method: Non-Probability Sample
Enrollment: 406 (Estimated)
Dates: Start 2025-08-22 (Estimated); Primary Completion 2026-01-20 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Comparison of PeDiAC Score and IDS Score for Predicting Difficult Intubation in Children Aged 0-5 Years | Immediately after tracheal intubation
  This outcome measure evaluates the effectiveness of two scoring systems-PeDiAC and Intubation Difficulty Scale (IDS)-in reflecting the difficulty of tracheal intubation in pediatric patients aged 0 to 5 years. Both scores will be calculated for each patient immediately after intubation. The correlation between each score and the actual intubation experience will be statistically analyzed to determine which scoring system better predicts intubation difficulty.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Bilkent City Hospital, Department Of Anesthesiology and Reanimation, Ankara, Turkey (Türkiye)